CLINICAL TRIAL: NCT01364558
Title: A Three-Period, Three-Treatment, Six-Sequence Randomized Crossover Study of the Bioavailability and Pharmacokinetics of Diazepam After Intranasal and Intravenous Administration to Healthy Volunteers",
Brief Title: A Study of Diazepam After Intranasal and Intravenous Administration to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Neurelis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1012M93599
Record Dates: First submitted 2011-05-20; First posted 2011-06-02 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diazepam Nasal Spray Suspension (Experimental): Diazepam Nasal Suspension - 10 mg
  Interventions: Drug: Diazepam
- Diazepam Nasal Spray Solution (Experimental): Diazepam Nasal Spray Solution - 10 mg
  Interventions: Drug: Diazepam
- Diazepam injection (Active Comparator): Diazepam injection IV - 5 mg
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — Diazepam will be administered as a 5 mg dose given IV. The two nasal formulations will be given as a 10 mg dose.
  Other Names: Brand names include: Valium, Diastat
  Arms: Diazepam Nasal Spray Solution; Diazepam Nasal Spray Suspension
Drug: Diazepam — IV diazepam will be given as a 5 mg dose. The two nasal formulations will be given as 10 mg doses.
  Other Names: Valium Injectable, Diastat Rectal Gel

SUMMARY:
The purpose of this clinical research study is to assess the bioavailability and pharmacokinetics of two formulations of diazepam after intranasal (nasal spray) and injectable diazepam after intravenous (I.V.) administration

DETAILED DESCRIPTION:
Diazepam is a medication that is used for the treatment of seizures. It was approved by the Food and Drug Administration (FDA) for use in the United States and is currently sold as Valium® tablets, Diazepam Injection and Diastat® rectal gel.

This study will evaluate two intranasal (nasal spray) formulations of diazepam which will be supplied by Neurelis, Inc. The purpose of this clinical research study is to assess the bioavailability and pharmacokinetics of two formulations of diazepam after intranasal (nasal spray) and injectable diazepam after intravenous (I.V.) administration. "Bioavailability" is a measure of how much drug is absorbed and present in the blood. "Pharmacokinetics" means to study the way a drug enters and leaves the blood and tissues over time

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 and 45 years (inclusive).
2. Written informed consent to participate in the study.
3. Body mass index (BMI) between 19 and 30 kg/m², inclusive.
4. Female subjects of childbearing potential, defined as not surgically sterile or at least two years (2) postmenopausal, must agree to use one of the following forms of contraception from three (3) months prior through 12 days following the last dose of study drug: hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), IUD, or vasectomized partner (six months minimum). Subjects must have used the same method for at least three (3) months prior to starting the study.
5. No clinically significant abnormal findings in the medical history, on the physical examination, electrocardiogram (ECG), or clinical laboratory results during Screening.
6. Subjects must agree to return to the study site for all study visits, including the three (3) confinement periods, and must be willing to comply with all required study procedures.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, severe seasonal or non seasonal allergies, nasal polyps or any nasal passage abnormality that could interfere with nasal spray administration, or any other condition which, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. A history of allergic or adverse responses to diazepam or any comparable or similar product.
3. Subjects who (for whatever reason) have been on an abnormal diet (such as one that severely restricts specific basic food groups [e.g., ketogenic diet], limits calories [e.g., fast], and/or requires the use of daily supplements as a substitute for the foods typically eaten at mealtimes), during the four (4) weeks preceding the study.
4. Subjects who donated blood or plasma within 30 days of the first dose of study drug.
5. Participation in a clinical trial within 30 days prior to the first dose of study drug. Participation in an observational (non interventional) study is not excluded as long as there are no scheduling conflicts with this study.
6. Inadequate or difficult venous access that may jeopardize the quality or timing of the PK samples.
7. Use of any over the counter (OTC) medication, including vitamins, within seven (7) days prior to the first dose of the study drug or during the study, unless approved by the Principal Investigator.
8. Use of any prescription medication, including benzodiazepines, within 14 days prior to the first dose of study drug or during the study, with the exception of hormonal contraceptives for women of childbearing potential, unless approved by the Principal Investigator.
9. Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study drug or during the study.
10. Smoking or use of tobacco products within six (6) months prior to the first dose of study drug or during the study.
11. Female subjects who are trying to conceive, are pregnant, or are lactating.
12. Positive serum pregnancy test at Screening or urine pregnancy test prior to each administration of study drug for all women, regardless of childbearing potential.
13. Positive blood screen for HIV, Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive urine screen for alcohol, drugs of abuse, or cotinine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cloyd, Pharm D., Principal Investigator — University of Minnesota
Locations (1):
- Prism Clinical Research Unit, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 24 subjects were given each formulation with a two week wash out period.
Groups:
- Diazepam Nasal Spray Suspension: Diazepam Nasal Spray Suspension
- Diazepam Nasal Spray Solution: Diazepam Nasal Spray Solution
- Diazepam Injection: Diazepam injection
Period: Dose One
Arm/Group | Diazepam Nasal Spray Suspension | Diazepam Nasal Spray Solution | Diazepam Injection
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Dose Two
Arm/Group | Diazepam Nasal Spray Suspension | Diazepam Nasal Spray Solution | Diazepam Injection
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Dose Three
Arm/Group | Diazepam Nasal Spray Suspension | Diazepam Nasal Spray Solution | Diazepam Injection
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diazepam Nasal Spray Suspension/Spray/Injection
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Absolute Bioavailability of Two Intranasal Diazepam Formulations.
Description: To calculate bioavailability we used the following formula:
  Area Under the Curve (Intranasal Spray)*100/Area Under the Curve (Intravenous Injection)
Time Frame: 2 days
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage of Bioavailability
Arm/Group | Diazepam Nasal Spray Suspension | Diazepam Nasal Spray Solution | Diazepam Injection
Number analyzed (Participants) | 24 | 24 | 24
Percentage of Bioavailability | 69 [64 to 75] | 96.82 [90 to 105] | 100 [100 to 100]

ADVERSE EVENTS:
Arm/Group | Diazepam Nasal Spray Suspension | Diazepam Nasal Spray Solution | Diazepam Injection
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 13/24 | 10/24 | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diazepam Nasal Spray Suspension (N=24) | Diazepam Nasal Spray Solution (N=24) | Diazepam Injection (N=24)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
General Disorders (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Nervous system disorders (Nervous system disorders) | 4 (4) | 3 (3) | 6 (6)
Respitory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes